CLINICAL TRIAL: NCT03962101
Title: A Multicenter, Open-label, Uncontrolled Clinical Trial to Confirm the Tolerability of OPC-61815 in Patients With Congestive Heart Failure Who Have Difficulty With or Are Incapable of Oral Intake
Brief Title: Safety Trial of OPC-61815 Injection in Patients With Congestive Heart Failure Who Have Difficulty With or Are Incapable of Oral Intake
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 263-102-00004; JapicCTI-194715 (Other: JapicCTI)
Record Dates: First submitted 2019-04-18; First posted 2019-05-23 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPC-61815 injection (Experimental): Intravenous administration of OPC-61815 at 8 mg or 16 mg once daily for a maximum of 5 days. Starting with 8mg, increase the dose to 16mg on Day 2 or Day 3, according to the dose escalation criteria.
  Interventions: Drug: OPC-61815 injection

INTERVENTIONS:
Drug: OPC-61815 injection — Intravenous administration of OPC-61815 at 8 mg or 16 mg once daily for a maximum of 5 days. Starting with 8mg, increase the dose to 16mg on Day 2 or Day 3, according to the dose escalation criteria.

SUMMARY:
To confirm the tolerability of intravenous administration of OPC-61815 at 8 or 16 mg once daily for a maximum of 5 days to CHF patients with volume overload despite having received diuretics (injection) other than vasopressin antagonists and who have difficulty with or are incapable of oral intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving loop diuretic injection at a dose equivalent to furosemide 20 mg/day or higher
* CHF patients in whom lower limb edema, pulmonary congestion, and/or jugular venous distension due to volume overload is present
* Patients who are judged by the investigator or subinvestigator to have difficulty or be incapable of oral intake, including patients who are judged by the investigator or subinvestigator to require nothing by mouth(NPO) management
* Patients who are currently hospitalized or who are capable of being hospitalized from the time of informed consent until the end of the treatment period
* Patients who are capable of giving informed consent

Exclusion Criteria:

* Patients who are on a ventricular assist device
* Patients who have difficulty with spontaneous respiration or who have been on tracheal intubation under sedative therapy
* Patients with severe disturbed consciousness (ie, coma or stupor)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Gifu Prefectural General Medical Center, Gifu, Japan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 subjects were administered investigational medicinal product (IMP): 38 subjects with dose maintained at 8 mg, and 7 subjects with dose increased to 16 mg. None of the subjects reduced the dose after the dose was increased to 16 mg. All 45 subjects received at least one dose of IMP and thus were included in the safety analysis set. Overall, 41 subjects completed the trial (34 of those subjects completed the trial early), and 4 subjects were discontinued from the trial.
Period: Overall Study
Arm/Group | OPC-61815 Injection
Started | 45
Completed | 41
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Not related to medical events | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: subjects who received at least one dose of IMP
Arm/Group | OPC-61815 Injection
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: "An AE is defined as any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an AE that leads to death, is life-threatening, results in persistent or significant disability/incapacity, requires in-patient or prolonged hospitalization, results in a congenital anomaly/birth defect, or any other important medical event which is medically significant.
  A TEAE is an AE that occurs only after a subject has received IMP.
Time Frame: From the start of IMP administration (Day 1) up to 15 days
Population: Safety Analysis Set: subjects who received at least one dose of IMP
Measure: Number; unit: percentage of participants
Arm/Group | OPC-61815 Injection
Number analyzed (Participants) | 45
percentage of participants | 77.8

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline (before IMP administration on Day 1) at time of final IMP administration (day after final IMP administration). A negative change from baseline indicates improvement.
Time Frame: Baseline, Day after final IMP administration
Population: Subjects with both baseline and evaluation of the given parameter at the specific visit.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | OPC-61815 Injection
Number analyzed (Participants) | 44
kg | -3.01 [-3.79 to -2.23]

3. Secondary Outcome: Improvement Rate for Lower Limb Edema
Description: The improvement rate was defined as the percentage of subjects in whom a symptom was present at baseline and then markedly improved or improved after IMP administration. Improvement category is a 4-point scale below:
  * Markedly improved
  * Improved
  * Unchanged
  * Deteriorated
Time Frame: Baseline, Day after final IMP administration
Population: Efficacy Analysis Set: subjects who received at least one dose of IMP and had at least one postbaseline dose efficacy measurement.
  "Overall Number of Participants Analyzed" = number of subjects with baseline symptoms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-61815 Injection
Number analyzed (Participants) | 38
percentage of participants | 73.7 [56.9 to 86.6]

4. Secondary Outcome: Improvement Rate for Pulmonary Congestion
Description: as for outcome 3
Time Frame: Baseline, Day after final IMP administration
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OPC-61815 Injection
Number analyzed (Participants) | 44
percentage of participants | 81.8 [67.3 to 91.8]

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the start of IMP administration up to 15 days
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Groups:
- OPC-61815 Injection Maintained at 8 mg: Intravenous administration of OPC-61815 at 8 mg once daily for a maximum of 5 days.
- OPC-61815 Injection Increased to 16 mg: Intravenous administration of OPC-61815 at 8 mg or 16 mg once daily for a maximum of 5 days. Starting with 8 mg, increase the dose to 16 mg on Day 2 and onward, according to the dose escalation criteria.
Arm/Group | OPC-61815 Injection Maintained at 8 mg | OPC-61815 Injection Increased to 16 mg
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/38 | 0/7
Other Adverse Events (participants affected / at risk) | 22/38 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection Maintained at 8 mg (N=38) | OPC-61815 Injection Increased to 16 mg (N=7)
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-61815 Injection Maintained at 8 mg (N=38) | OPC-61815 Injection Increased to 16 mg (N=7)
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 11 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Injection site inflammation (General disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0
Urinary tract infection (Infections and infestations) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Delirium (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Phlebitis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03962101/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03962101/SAP_001.pdf